CLINICAL TRIAL: NCT01399684
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of MEGF0444A Dosed to Progression in Combination With Bevacizumab and FOLFOX in Patients With Previously Untreated Metastatic Colorectal Cancer
Brief Title: A Study Evaluating the Efficacy and Safety of MEGF0444A Dosed to Progression in Combination With Bevacizumab and mFOLFOX-6 in Participants With Previously Untreated Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEF4982g; GO27812 (Other: Hoffmann-La Roche); 2011-001867-28 (EudraCT Number)
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Bevacizumab; Leucovorin; parsatuzumab; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- MEGF0444A + mFOLFOX-6 + Bevacizumab (Experimental): Participants will receive MEGF0444A + mFOLFOX-6 (oxaliplatin, folinic acid, and 5-fluorouracil) regimen + bevacizumab. Participants will receive oxaliplatin for up to 8 cycles (Cycle = 14 days) and 5-fluorouracil, folinic acid, bevacizumab and MEGF0444A will be administered until disease progression or unacceptable toxicity for a maximum of up to 52 cycles.
  Interventions: Drug: 5-Fluorouracil; Drug: Bevacizumab; Drug: Folinic acid; Drug: MEGF0444A; Drug: Oxaliplatin
- Placebo + mFOLFOX-6 + Bevacizumab (Placebo Comparator): Participants will receive MEGF0444A matching placebo + mFOLFOX-6 regimen + bevacizumab. Participants will receive oxaliplatin for up to 8 cycles and 5-fluorouracil, folinic acid, bevacizumab and placebo will be administered until disease progression or unacceptable toxicity for a maximum of up to 52 cycles.
  Interventions: Drug: 5-Fluorouracil; Drug: Bevacizumab; Drug: Folinic acid; Drug: Oxaliplatin; Drug: Placebo

INTERVENTIONS:
Drug: 5-Fluorouracil — Participants will receive 5-fluorouracil 400 milligrams per squared meter (mg/m^2) intravenous (IV) bolus and then 2400 mg/m^2 as a continuous IV infusion over 46-48 hours on Day 1 of every cycle until disease progression, unacceptable toxicity or at the maximum of 52 cycles, whichever occurs first.
Drug: Bevacizumab — Participants will be administered bevacizumab at a dose of 5 milligrams per kilogram (mg/kg) every 14 days until disease progression or unacceptable toxicity, for a maximum of 52 cycles, whichever occurs first.
Drug: Folinic acid — Participants will receive folinic acid 400 mg/m^2 IV infusion over 2 hours on Day 1 of every cycle until disease progression, unacceptable toxicity or at the maximum of 52 cycles, whichever occurs first.
Drug: MEGF0444A — Participants will be administered MEGF0444A at a fixed dose of 400 milligrams (mg) IV on Day 1 of Cycle 1, followed by subsequent doses of 400 mg every 14 days until disease progression or unacceptable toxicity, for a maximum of 52 cycles, whichever occurs first.
  Arms: MEGF0444A + mFOLFOX-6 + Bevacizumab
Drug: Oxaliplatin — Participants will receive oxaliplatin 85 mg/m^2 IV infusion over 90 minutes on Day 1 of every cycle for a maximum of 8 cycles.
Drug: Placebo — Participants will be administered MEGF0444A matching placebo every 14 days until disease progression, unacceptable toxicity or at the maximum of 52 cycles, whichever occurs first.
  Arms: Placebo + mFOLFOX-6 + Bevacizumab

SUMMARY:
This is a Phase II, multicenter, randomized, double-blind, placebo-controlled trial designed to estimate the efficacy of MEGF0444A treatment to disease progression, combined with oxaliplatin + folinic acid + 5-Fluorouracil (mFOLFOX-6) + bevacizumab therapy in participants with metastatic colorectal cancer (CRC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed CRC not amenable to potentially curative resection with at least one measurable metastatic lesion, as defined by RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic and end organ function
* For female participants of childbearing potential and male participants with partners of childbearing potential, agreement to use a highly effective form of contraception and to continue its use for 6 months after the last dose of study treatment
* Negative serum pregnancy test within 7 days prior to starting study treatment in premenopausal women and women less than (<) 2 years after the onset of menopause

Exclusion Criteria:

Disease-specific exclusions

* Any prior systemic therapy (including chemotherapy, antibody therapy, tyrosine kinase inhibitors, radiotherapy, immunotherapy, hormonal therapy or investigational therapy) before Day 1 of Cycle 1 for treatment of CRC General Medical Exclusions
* Malignancies other than CRC within 5 years prior to randomization, except for those with a negligible risk of metastasis or death
* Radiotherapy to any site for any reason within 28 days prior to Day 1 of Cycle 1
* Clinically detectable third-space fluid collections that cannot be controlled by drainage or other procedures prior to study entry
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to Day 1 of Cycle 1
* Lactating women
* Clinically suspected or confirmed central nervous system (CNS) metastases or carcinomatous meningitis
* Active infection requiring IV antibiotics
* Active autoimmune disease that is not controlled by nonsteroidal anti-inflammatory drugs, inhaled corticosteroids, or the equivalent of less than or equal to (</=) 10 milligrams per day (mg/day) prednisone
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, or cirrhosis
* Sensory peripheral neuropathy greater than or equal to (>/=) Grade 2 Bevacizumab-Specific Exclusions
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of bevacizumab or an investigational drug or that may affect the interpretation of the results or render the participant at high risk for treatment complications
* Inadequately controlled hypertension
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Class II or greater congestive heart failure (CHF)
* History of myocardial infarction or unstable angina within 6 months prior to Day 1
* History of stroke or transient ischemic attack (TIA) within 6 months prior to Day 1
* Significant vascular disease within 6 months prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy
* Current or recent (within 10 days of first dose of study treatment) use of aspirin or treatment with dipyramidole, ticlopidine, clopidogrel, and cilostazol
* Current or recent (within 10 days prior to study treatment start) use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purpose
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1, or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
* History of abdominal or tracheo-oesophageal fistula or gastrointestinal (GI) perforation within 6 months prior to Day 1
* Clinical signs or symptoms of GI obstruction or a requirement for routine parenteral hydration, parenteral nutrition, or tube feeding
* Evidence of abdominal free air not explained by paracentesis or recent surgical procedure
* Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture 5-Fluorouracil-Specific Exclusion
* Known dihydropyrimidine dehydrogenase deficiency or thymidylate synthase gene polymorphism predisposing the participant for 5-fluorouracil toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2011-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival Based on Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1 as Determined by the Investigator | Screening up to disease progression or death due to any cause, whichever occurs first (assessed every 8-9 weeks after Cycle 1 Day 1 up to approximately 27 months overall)

SECONDARY OUTCOMES:
Percentage of Participants with Objective Response (Complete Response [CR] or Partial Response [PR] Based on RECIST v 1.1 as Determined by the Investigator | Screening up to disease progression or death due to any cause, whichever occurs first (assessed every 8 -9 weeks after Cycle 1 Day 1 up to approximately 27 months overall)
Duration of Response Based on RECIST v 1.1 as Determined by the Investigator | Screening up to disease progression or death due to any cause, whichever occurs first (assessed every 8 -9 weeks after Cycle 1 Day 1 up to approximately 27 months overall)
Overall Survival (OS) | Screening until death (up to approximately 27 months overall)
Percentage of Participants with Adverse Events | Up to approximately 27 months overall
Maximum Serum Concentration (Cmax) of MEGF0444A | Prior to the first infusion (first infusion being MEGF0444A administration), immediately after end of bevacizumab infusion on Day 1 of Cycles 1, 2; prior to first infusion on Day 1 of Cycles 3 and 8; at study drug discontinuation visit (up to 24 months)
Minimum Serum Concentration (Cmin) of MEGF0444A | Prior to the first infusion (first infusion being MEGF0444A administration), immediately after end of bevacizumab infusion on Day 1 of Cycles 1, 2; prior to first infusion on Day 1 of Cycles 3 and 8; at study drug discontinuation visit (up to 24 months)
Cmax of Bevacizumab | Prior to the first infusion (first infusion being MEGF0444A administration), immediately after end of bevacizumab infusion on Day 1 of Cycles 1, 2
Cmin of Bevacizumab | Prior to the first infusion (first infusion being MEGF0444A administration), immediately after end of bevacizumab infusion on Day 1 of Cycles 1, 2
Plasma Concentration of 5-Fluorouracil | Prior to the first infusion (first infusion being MEGF0444A administration), immediately after end of 5-fluorouracil bolus, 2 hours after end of 5-fluorouracil bolus, 12-24 hours after end of 5-fluorouracil bolus on Day 1 of Cycles 1, 2
Plasma Concentration of Oxaliplatin | Prior to the first infusion (first infusion being MEGF0444A administration), 5-10 minutes before end of oxaliplatin infusion, 2 hours after end of 5-fluorouracil bolus, 12-24 hours after end of 5-fluorouracil bolus on Day 1 of Cycles 1, 2
Percentage of Participants with Anti-Therapeutic Antibodies (ATAs) to MEGF0444A | Pre-dose (within 1 hour before infusion start) on Day 1 of Cycles 1, 3 and 8, (cycle length = 14 days), at study drug discontinuation visit (up to 24 months)
Change From Baseline in ATAs Levels of MEGF0444A | Pre-dose (within 1 hour before infusion start) on Day 1 of Cycles 1, 3 and 8, (cycle length = 14 days), at study drug discontinuation visit (up to 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Ina Rhee, M.D., Ph.D., Study Director — Genentech, Inc.
Locations (36):
- United States (21):
  - Birmingham, Alabama
  - Scottsdale, Arizona
  - Bakersfield, California
  - Fullerton, California
  - Los Angeles, California
  - Pasadena, California
  - San Luis Obispo, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Ocala, Florida
  - Port Saint Lucie, Florida
  - Lawrenceville, Georgia
  - Marietta, Georgia
  - Harvey, Illinois
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Rochester, Minnesota
  - Las Vegas, Nevada
  - Durham, North Carolina
  - Philadelphia, Pennsylvania
- Australia (5):
  - South Brisbane, Queensland
  - Woodville South, South Australia
  - Footscray, Victoria
  - Heidelberg, Victoria
  - Melbourne, Victoria
- Belgium (2):
  - Brussels
  - Leuven
- Poland (4):
  - Gdansk
  - Krakow
  - Poznan
  - Warsaw
- Spain (4):
  - Barcelona, Barcelona
  - Santander, Cantabria
  - Seville, Sevilla
  - Valencia, Valencia

REFERENCES:
- [Derived] Garcia-Carbonero R, van Cutsem E, Rivera F, Jassem J, Gore I Jr, Tebbutt N, Braiteh F, Argiles G, Wainberg ZA, Funke R, Anderson M, McCall B, Stroh M, Wakshull E, Hegde P, Ye W, Chen D, Chang I, Rhee I, Hurwitz H. Randomized Phase II Trial of Parsatuzumab (Anti-EGFL7) or Placebo in Combination with FOLFOX and Bevacizumab for First-Line Metastatic Colorectal Cancer. Oncologist. 2017 Apr;22(4):375-e30. doi: 10.1634/theoncologist.2016-0133. Epub 2017 Mar 8. PMID 28275117